CLINICAL TRIAL: NCT00807690
Title: Treatment of Vitiligo With Narrowband UVB (TL01) Combined With Tacrolimus (0.1%) Versus Placebo Ointment, a Randomized Right/Left Double Blind Comparative Study
Brief Title: Vitiligo Treated With TL01 Combined With Tacrolimus Ointment Versus Placebo
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Eli Johanne Nordal/senior consultant, Rikshospitalet HF
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 182-04066
Record Dates: First submitted 2008-12-11; First posted 2008-12-12 (Estimated); Last update posted 2008-12-12 (Estimated); Status verified 2008-12

CONDITIONS: Vitiligo
Keywords: vitiligo; tacrolimus ointment 0.1%; narrowband UVB (TL01)
MeSH Terms: conditions — Vitiligo

INTERVENTIONS:
Drug: Tacrolimus ointment — Tacrolimus ointment 0.1%every night for at least 3 months, half body side

SUMMARY:
BACKGROUND Vitiligo is a common, often distressing condition. Many of the patients do not achieve sufficient effect from what is regarded as the treatment of choice at present, narrow band(NB)UVB(Tl01). There are reports on some patients partly successfully treated with Tacrolimus ointment.

AIM OF THE STUDY We want to study whether Tacrolimus ointment may give an additive effect on symmetric vitiligo in combination with NB-UVB.

METHODS This is a double blind left/right comparative study with 6 months treatment time. Patients are treated with whole body NB-UVB x 2 or x 3 weekly, in addition to Tacrolimus ointment versus placebo every night on affected half body sites. To measure effects we use photodocumentation in addition to morphometric registration of symmetric target lesions every 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged at least 18 years with a stable, symmetric vitiligo

Exclusion Criteria:

* Patients with segmental vitiligo, aged < 18 years, known hypersensitivity to Tacrolimus, pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-11; Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eli Johanne Nordal, MD, Principal Investigator — Rikshospitalet HF, Dept. of Dermatology